CLINICAL TRIAL: NCT04000594
Title: An Open-Label Adaptive Multiple-Dose Study to Investigate the Pharmacokinetics and Pharmacodynamics of RO7234292 in CSF and Plasma, and Safety and Tolerability Following Intrathecal Administration in Patients With Huntington's Disease
Brief Title: A Study to Investigate the Pharmacokinetics and Pharmacodynamics of RO7234292 (RG6042) in CSF and Plasma, and Safety and Tolerability Following Intrathecal Administration in Patients With Huntington's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP40410; GEN-PEAK (Other: Hoffmann-La Roche)
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Huntingtons Disease
MeSH Terms: conditions — Chorea | interventions — tominersen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose level 1 of RO7234292 (RG6042) (Experimental): Participants will receive dose level 1 of RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
  Interventions: Drug: RO7234292 (RG6042)
- Dose level 2 of RO7234292 (RG6042) (Experimental): Participants will receive dose level 2 of RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
  Interventions: Drug: RO7234292 (RG6042)
- Dose level 3 of RO7234292 (RG6042) (Experimental): Participants will receive dose level 3 of RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
  Interventions: Drug: RO7234292 (RG6042)

INTERVENTIONS:
Drug: RO7234292 (RG6042) — RO7234292 (RG6042) will be administered in two IT doses of the same dose level at an interval of 28 days during the treatment period (Day 1 and Day 29). Each dose of RO7234292 (RG6042) will be administered as a single IT bolus injection.
  Other Names: Tominersen

SUMMARY:
Study BP40410 is an open-label, adaptive multiple-dose clinical study designed to characterize the PK of RO7234292 (RG6042) in plasma and CSF as well as the acute time course and recovery profile of CSF mHTT lowering in response to RO7234292 (RG6042) treatment after intrathecal (IT) administration of RO7234292 (RG6042) to patients with manifest Hungtington's disease (HD).

ELIGIBILITY:
Inclusion Criteria:

* Manifest HD diagnosis
* Independence Scale score of >=70.
* Genetically confirmed disease by direct deoxyribonucleic acid testing with a cytosine, adenine, and guanine base sequence found in DNA which is translated into glutamine (CAG) age product (CAP) score > 400.
* Ability to read the words "red," "blue," and "green" in the patient's native language.
* Ability to walk unassisted without a cane or walker and move about without a wheelchair on a daily basis as reviewed at screening and baseline visit.
* Ability to undergo and tolerate MRI scans.

Exclusion Criteria:

* History of attempted suicide or suicidal ideation with plan (i.e., active suicidal ideation) that required hospital visit and/or change in level of care within 12 months prior to screening.
* Current active psychosis, confusional state, or violent behavior.
* Any serious medical condition or clinically significant laboratory, vital signs, or ECG abnormalities at screening that, in the Investigator's judgment, precludes the patient's safe participation in and completion of the study.
* Clinical diagnosis of chronic migraines or history of low pressure headache after lumbar puncture requiring hospitalization or blood patch.
* Treatment with investigational therapy within 4 weeks prior to screening or 5 drug elimination half-lives of investigational therapy, whichever is longer.
* Concurrent or planned concurrent participation in any interventional clinical study, including explicit pharmacological and non-pharmacological interventions. Observational studies are acceptable.
* Unable or unsafe to perform lumbar puncture on the patient.
* Previous lumbar surgery that is likely, in the opinion of the Investigator or surgical team, to make IT catheter insertion or IT injection unduly difficult or hazardous.
* Poor peripheral venous access.
* Scoliosis or spinal deformity making IT injection not feasible in the outpatient setting.
* Preexisting intra-axial or extra-axial lesions as assessed by a centrally read MRI scan during the screening period.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Centre For Human Drug Research; Research, Leiden, Netherlands
- United Kingdom (2):
  - Leonard Wolfson Experimental Neurology Centre, London
  - Manchester University NHS Foundation Trust (MFT), Manchester

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 of RO7234292 (RG6042): Participants received dose level 1 of 30 mg RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
- Dose Level 2 of RO7234292 (RG6042): Participants received dose level 2 of 60 mg RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
- Dose Level 3 of RO7234292 (RG6042): Participants received dose level 3 of 120 mg RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
Period: Overall Study
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Started | 4 | 4 | 4
Completed | 3 | 4 | 4
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (12.2) | 45.8 (10.9) | 53.8 (6.9) | 47.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 3 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of RO7234292 in CSF (Cerebrospinal Fluid)
Description: NA represents: insufficient number of participants with events.
Time Frame: Day 1, 2, 3, 4, 29, 43, 71, 127, and follow-up visit (6 months after last study drug administration)
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  Day 1 2 hour: number analyzed (Participants) | 4 | 3 | 4
  Day 1 2 hour | 197000 (71400) | 372000 (132000) | 933000 (349000)
  Day 2 24 hour: number analyzed (Participants) | 4 | 3 | 4
  Day 2 24 hour | 6220 (6270) | 30200 (17300) | 41100 (20000)
  Day 3 48 hour: number analyzed (Participants) | 4 | 3 | 4
  Day 3 48 hour | 888 (1510) | 4540 (3510) | 6880 (4830)
  Day 4 72 hour: number analyzed (Participants) | 0 | 1 | 4
  Day 4 72 hour |  | NA (NA) — insufficient number of patients with available measures | 1270 (1070)
  Day 29: number analyzed (Participants) | 3 | 3 | 3
  Day 29 | 1.08 (0.773) | 1.51 (0.757) | 2.64 (0.572)
  Day 43: number analyzed (Participants) | 3 | 3 | 3
  Day 43 | 2.81 (0.906) | 3.97 (1.85) | 6.79 (1.15)
  Day 71: number analyzed (Participants) | 3 | 2 | 3
  Day 71 | 1.08 (0.459) | 1.78 (0.0919) | 2.92 (0.570)
  Day 127: number analyzed (Participants) | 3 | 2 | 1
  Day 127 | 0.329 (0.129) | 0.416 (0.0361) | NA (NA) — insufficient number of patients with available measures
  Follow-up: number analyzed (Participants) | 2 | 2 | 0
  Follow-up | NA (NA) — insufficient number of patients with available measures | NA (NA) — insufficient number of patients with available measures |

2. Primary Outcome: Concentrations of RO7234292 in Plasma
Description: NA represents:insufficient number of participants with events
Time Frame: Day 1, 2, 3, 4, 5, 28, 29, 30, 43, 71, 127, and follow-up visit (6 months after last study drug administration)
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  Day 1 1 hour | 209 (173) | 709 (765) | 941 (625)
  Day 2 24 hour | 30.5 (31.1) | 709 (765) | 104 (84.6)
  Day 3 48 hour | 2.66 (4.05) | 5.87 (5.36) | 12.8 (5.73)
  Day 4 72 hour | 0.480 (0.192) | 1.76 (1.25) | 4.20 (2.11)
  Day 28: number analyzed (Participants) | 2 | 3 | 3
  Day 28 | NA (NA) — insufficient number of patients with available measures | 0.119 (0.0273) | 0.316 (0.114)
  Day 29: number analyzed (Participants) | 3 | 4 | 3
  Day 29 | 0.142 (0.143) | 0.135 (0.132) | 0.292 (0.0887)
  Day 30: number analyzed (Participants) | 3 | 3 | 3
  Day 30 | 46.4 (27.1) | 103 (52.0) | 317 (57.6)
  Day 43: number analyzed (Participants) | 3 | 3 | 4
  Day 43 | 0.249 (0.140) | 0.356 (0.195) | 0.983 (0.401)
  Day 71: number analyzed (Participants) | 1 | 1 | 3
  Day 71 | NA (NA) — insufficient number of patients with available measures | NA (NA) — insufficient number of patients with available measures | 0.983 (0.401)
  Day 127: number analyzed (Participants) | 0 | 1 | 0
  Day 127 |  | NA — insufficient number of patients with available measures |
  Follow-up visit: number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: mHTT (Mutant Huntingtin) Concentration in CSF
Description: CSF Mutant Huntingtin Protein (fmol/L) values at time point visits are reported.
Time Frame: Days 1, 2, 3, 29, 43, 71, 127 and follow-up visit (6 months after last study drug administration)
Population: PK Population
Measure: Mean (Standard Deviation); unit: fmol/L
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
fmol/L
  Day 1 4H: number analyzed (Participants) | 4 | 3 | 4
  Day 1 4H | 177.78 (92.81) | 130.35 (40.16) | 99.02 (50.65)
  Day 2 24H: number analyzed (Participants) | 2 | 2 | 4
  Day 2 24H | 204.39 (180.26) | 81.74 (22.38) | 127.39 (42.40)
  Day 3 48H: number analyzed (Participants) | 3 | 3 | 4
  Day 3 48H | 325.18 (215.71) | 190.85 (161.19) | 176.59 (125.52)
  Day 29 Pre-dose: number analyzed (Participants) | 3 | 2 | 3
  Day 29 Pre-dose | 107.46 (85.36) | 91.53 (20.65) | 55.62 (16.70)
  Day 43: number analyzed (Participants) | 3 | 2 | 3
  Day 43 | 83.75 (41.84) | 66.07 (1.08) | 68.92 (21.89)
  Day 71: number analyzed (Participants) | 3 | 2 | 3
  Day 71 | 138.25 (127.63) | 74.86 (14.38) | 49.24 (12.50)
  Day 127: number analyzed (Participants) | 3 | 2 | 3
  Day 127 | 127.80 (112.79) | 81.05 (21.84) | 41.55 (10.96)
  Follow-Up: number analyzed (Participants) | 3 | 3 | 4
  Follow-Up | 132.13 (115.59) | 68.77 (24.49) | 61.55 (8.84)

4. Secondary Outcome: Percentage of Participants With Adverse Events According to NCI-CTCAE Grading System
Description: Severity levels levels: 1 = mild; 2 = moderate; 3 = severe used according to NCI-CTCAE grading system.
  Percentage of participants with 1-3 levels of severities are reported.
Time Frame: Up to 6 months
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
Percentage of Participants
  Any Adverse Events Level 1 | 50 | 0 | 50.0
  Any Adverse Events Level 2 | 25 | 75 | 25.0
  Any Adverse Events Level 3 | 25 | 25 | 25.0
  Injury, poisoning and procedural complications Level 1 | 50 | 25 | 50
  Injury, poisoning and procedural complications Level 2 | 50 | 50 | 25
  Injury, poisoning and procedural complications Level 3 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders Level 1 | 75 | 50 | 50
  Musculoskeletal and connective tissue disorders Level 2 | 25 | 0 | 25
  Musculoskeletal and connective tissue disorders Level 3 | 0 | 25 | 0
  Nervous system disorders Level 1 | 25.0 | 25.0 | 75
  Nervous system disorders Level 2 | 0 | 25 | 0
  Nervous system disorders Level 3 | 25 | 0 | 0
  General disorders and administration site conditions Level 1 | 0 | 25.0 | 0
  General disorders and administration site conditions Level 2 | 25 | 25 | 25
  General disorders and administration site conditions Level 3 | 0 | 0 | 25
  Infections and infestations Level 1 | 0 | 0 | 25
  Infections and infestations Level 2 | 25 | 25 | 0
  Infections and infestations Level 3 | 0 | 25 | 25
  Gastrointestinal disorders Level 1 | 25 | 0 | 50
  Gastrointestinal disorders Level 2 | 0 | 25 | 0
  Gastrointestinal disorders Level 3 | 0 | 0 | 0
  Ear and labyrinth disorders Level 1 | 25 | 0 | 0
  Ear and labyrinth disorders Level 2 | 0 | 0 | 0
  Ear and labyrinth disorders Level 3 | 0 | 0 | 0
  Investigations Level 1 | 0 | 0 | 0
  Investigations Level 2 | 0 | 25 | 0
  Investigations Level 3 | 0 | 0 | 0
  Metabolism and nutrition disorders Leve 1 | 0 | 0 | 25
  Metabolism and nutrition disorders Leve 2 | 0 | 0 | 0
  Metabolism and nutrition disorders Leve 3 | 0 | 0 | 0
  Psychiatric disorders Level 1 | 0 | 25 | 0
  Psychiatric disorders Level 2 | 0 | 0 | 0
  Psychiatric disorders Level 3 | 0 | 0 | 0
  Reproductive system and breast disorders Level 1 | 0 | 0 | 0
  Reproductive system and breast disorders Level 2 | 25 | 0 | 0
  Reproductive system and breast disorders Level 3 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders Level 1 | 0 | 0 | 25
  Respiratory, thoracic and mediastinal disorders Level 2 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders Level 3 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders Level 1 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders Level 2 | 0 | 0 | 25
  Skin and subcutaneous tissue disorders Level 3 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Suicidal Ideation or Behavior, as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a structured tool to assess suicidal ideation and behavior.
  Four constructs are measured: severity of ideation, intensity of ideation, behavior, and lethality of actual suicide attempts. Binary (yes/no) data are collected for 10 categories, and composite endpoints based on the categories are followed over time to monitor patient safety. Scores 1-10 is used, 1 being less and to 10 being severity increasing.
  Only one time frame was used per score category: from screening to follow-up visit.
Time Frame: From Screening Day Up To Follow-up Visit (6 months after the last Dosing Day-Day 127)
Population: ITT
Measure: Number; unit: Percentage
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
Percentage
  Suicidal Ideation (score 1-5) -Wish to Be Dead | 0 | 25 | 0
  Suicidal Ideation (score 1-5) -Non-specific Active Suicidal Thoughts | 0 | 0 | 0
  -Active Suicidal Ideation with Any Suicidal Ideation (score 1-5) -Methods (Not Plan) without Intent | 0 | 0 | 0
  Suicidal Ideation (score 1-5) -Intent to Act, without Plan Active Suicidal Ideation | 0 | 0 | 0
  Suicidal Ideation (score 1-5) -Active Suicidal Ideation with Specific Plan and Intent | 0 | 0 | 0
  Suicidal Behavior (6-10) -Preparatory Acts or Behavior | 0 | 0 | 0
  Suicidal Behavior (6-10) -Aborted Attempt | 0 | 0 | 0
  Suicidal Behavior (6-10) -Interrupted Attempt | 0 | 0 | 0
  Suicidal Behavior (6-10) -Non-fatal Suicide Attempt | 0 | 0 | 0
  Suicidal Behavior (6-10) -Completed Suicide | 0 | 0 | 0
  Suicidal Behavior (6-10) -Self-injurious Behavior without Suicidal Intent | 0 | 0 | 0

6. Secondary Outcome: Incidence of Anti-Drug Antibodies (ADAs)
Description: Percentage of participants who have negative or positive anti-drug antibody affects are reported.
Time Frame: Day 1, Day 28, and follow-up visit (6 months after last study drug administration)
Population: Safety Population
Measure: Number; unit: Percentage
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
Percentage
  Baseline Day 1 Total Negative: number analyzed (Participants) | 3 | 4 | 4
  Baseline Day 1 Total Negative | 100 | 100 | 100
  Day 28 Total Negative: number analyzed (Participants) | 3 | 4 | 3
  Day 28 Total Negative | 100 | 100 | 100
  Follow-up Total Negative: number analyzed (Participants) | 3 | 4 | 4
  Follow-up Total Negative | 100 | 100 | 100

7. Secondary Outcome: Titer and Antibody Subtype, Determined if ADAs Are Identified
Description: The data cannot be reported and the outcome measure is not applicable as no ADA sample was positive. As no ADA, titer and subtype could not be identified
Time Frame: Day 1, Day 28, and follow-up visit (6 months after last study drug administration)
Population: No data evaluable participants
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Amount of RO7234292 in Urine Ae (Micrograms)
Time Frame: Up to 72 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms
Arm/Group | Dose Level 1 of RO7234292 (RG6042) | Dose Level 2 of RO7234292 (RG6042) | Dose Level 3 of RO7234292 (RG6042)
Number analyzed (Participants) | 4 | 4 | 4
micrograms | 236.0 (78.0) | 207.0 (131.0) | 1650.0 (53.0)

ADVERSE EVENTS:
Time Frame: The 2nd dose (last dose) of study drug on Day 29 and the last follow-up visit was 6 months after the last dose.
Groups:
- 30 MG RG6042: Participants received dose level 1 of 30 mg RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
- 60 MG RG6042: Participants will receive dose level 2 of 60 mg RO7234292 (RG6042) intrathecally on Day 1 and Day 29
- 120 MG RG6042: Participants will receive dose level 3 of 120 mg RO7234292 (RG6042) intrathecally on Day 1 and Day 29.
Arm/Group | 30 MG RG6042 | 60 MG RG6042 | 120 MG RG6042
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 MG RG6042 (N=4) | 60 MG RG6042 (N=4) | 120 MG RG6042 (N=4)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 MG RG6042 (N=4) | 60 MG RG6042 (N=4) | 120 MG RG6042 (N=4)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device site vesicles (General disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (4)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04000594/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04000594/SAP_001.pdf